CLINICAL TRIAL: NCT06185023
Title: Exercising Language: Behavioral and Neurophysiological Changes After High-intensity Exercise Training in Post-stroke Aphasia
Brief Title: Effects of High-intensity Exercise Training on Physical Fitness, Cognition, Language in Post-stroke Aphasia
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Collaborators: University of California, San Francisco (Other); University of San Francisco (Other); California State University, East Bay (Other)
Responsible Party: Principal Investigator, Maria Ivanova, Assistant Professional Researcher, University of California, Berkeley
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 056427-002
Record Dates: First submitted 2023-12-14; First posted 2023-12-29 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Aphasia, Acquired; Aphasia; Aphasia, Fluent; Aphasia Non Fluent
Keywords: aphasia; physical exercise; high intensity interval training; cognition; physical fitness; balance
MeSH Terms: conditions — Aphasia; Aphasia, Wernicke; Aphasia, Broca; Motor Activity

STUDY DESIGN:
Intervention Model Description: As this is a feasibility study, participants can choose to participate in just one or both types of physical exercise interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low-intensity physical exercise (Active Comparator): The participants will participate in a low-intensity non-aerobic exercise program for 2 weeks.
  Interventions: Behavioral: Low-intensity physical exercise
- High-intensity physical exercise (Experimental): The participants will take part in a high-intensity Aphasia Physical EXercise (APEX) intervention designed specifically for individuals with chronic post-stroke aphasia for 8 weeks.
  Interventions: Behavioral: High-intensity physical exercise
- High-intensity physical exercise - remote (Experimental): The participants will take part in a high-intensity Aphasia Physical EXercise (APEX) intervention designed specifically for individuals with chronic post-stroke aphasia for 4 weeks. The first week will be delivered in-person, while weeks 2-4 will be delivered remotely via live Zoom classes.
  Interventions: Behavioral: High-intensity physical exercise

INTERVENTIONS:
Behavioral: Low-intensity physical exercise — As an active control intervention, a low-intensity non-aerobic exercise program was selected that mirrors more closely the standard-of-care physical therapy currently provided to stroke patients. This control intervention will offer the same level of participant involvement and type of exercises, but without the intensity element, i.e., it will not incorporate the cardiovascular and the strengthening components.
  Arms: Low-intensity physical exercise
Behavioral: High-intensity physical exercise — We have developed a new exercise program specifically designed for individuals with post-stroke aphasia, Aphasia Physical EXercise (APEX), to provide a safe, stroke- and aphasia-friendly physical exercise intervention to achieve optimal physical fitness and cognitive/language gains. This intervention, based on published research and clinical practice recommendations, is a high-intensity interval training full-body workout optimized to accommodate the range of motor abilities and general deconditioning observed in stroke survivors.
  Arms: High-intensity physical exercise; High-intensity physical exercise - remote

SUMMARY:
The goal of this clinical trial is to establish the feasibility and fidelity of a high-intensity exercise program for individuals with post-stroke aphasia. The main questions it aims to answer are:

* Is it feasible for stroke survivors with aphasia to participate in a long in-person physical exercise program?
* Does participation in a physical exercise program lead to physical fitness, cognitive, language and/or psychological changes?

Participants can take part in two different physical exercise interventions:

* Low intensity intervention (control intervention);
* High-intensity physical exercise intervention (target intervention).

ELIGIBILITY:
Inclusion Criteria:

* aphasia following single or multiple ischemic or hemorrhagic stroke;
* at least 6 months from the last stroke;
* proficient in English before the stroke;
* at least 8 years of education;
* between the ages of 18 and 80;
* independent with ambulation without a device (single-point cane accepted);
* medically stable with no contraindications to participate in regular physical exercise as determined by the patient's own primary care provider or other treating provider.

Exclusion Criteria:

* prior history of dementia, neurologic illness (other than stroke), or substance abuse;
* significant visual or hearing disabilities (e.g., neglect, uncorrected visual or hearing loss) that interfere with testing;
* per self-report uncontrolled cardiorespiratory and/or metabolic disorders incompatible with exercise.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-12-12 (Actual); Primary Completion 2025-09-12 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change on the Western Aphasia Battery (WAB) - Aphasia Quotient | Baseline and immediately after the intervention (3rd week for the low-intensity arm and 9th week for the high-intensity arm)
  The Aphasia Quotient from the Western Aphasia Battery (a standardized language test) measures overall severity of language impairment in aphasia and ranges from 0 to 100, with lower scores indicative of more severe aphasia.

SECONDARY OUTCOMES:
Changes in Maximal Aerobic Capacity | Baseline and immediately after the intervention (3rd week for the low-intensity arm and 9th week for the high-intensity arm)
  This is a measure of cardiorespiratory and metabolic fitness. Maximal Aerobic Capacity (VO2 Max) is the ability of the body to utilize oxygen to produce energy and is measured via a graded exercise test until volitional fatigue, while measuring consumption of oxygen with a computerized metabolic system. Typically measured on a treadmill, VO2 Max has also been found to be accurately and safely measured in stroke survivors on a recumbent stepper, which will be used in this study. A good VO2max varies greatly depending on age, and for older participants is typically between 30-40 ml/kg/min (higher values indicate greater fitness).
Attendance | After the intervention (3rd week for the control intervention and 9th week for the experimental intervention)
  Total number of physical exercise classes attended during the intervention.
Change on the 30-second chair stands | Baseline and immediately after the intervention (3rd week for the low-intensity arm and 9th week for the high-intensity arm)
  The number of full stands from a seated position that can be completed in 30 seconds with arms folded across the chest.
Change on the 2-minute Step Test | Baseline and immediately after the intervention (3rd week for the low-intensity arm and 9th week for the high-intensity arm)
  The number of knee raises completed in 2 minutes, raising each knee to a point midway between the patella (kneecap) and iliac crest (top hip bone).
Change on the Timed Up-and-Go Test | Baseline and immediately after the intervention (3rd week for the low-intensity arm and 9th week for the high-intensity arm)
  The number of seconds it takes to get up from a seated position, walk 3 m, turn, and return to a seated position.
Change on the Functional Reach Test | Baseline and immediately after the intervention (3rd week for the low-intensity arm and 9th week for the high-intensity arm)
  The number of inches reached forward with each arm with feet flat on the floor at hip width.
Change in Gait Speed | Baseline and immediately after the intervention (3rd week for the low-intensity arm and 9th week for the high-intensity arm)
  The speed in meters per second for the middle 6 m of the 10 m walkway.

OTHER OUTCOMES:
Change on the Philadelphia Naming Test (PNT) | Baseline and immediately after the intervention (3rd week for the low-intensity arm and 9th week for the high-intensity arm)
  Aphasia naming test to assess word retrieval abilities. The score ranges from 0 to 100, with a higher score indicating greater naming ability.
Change on the Curtiss-Yamada Comprehensive Language Evaluation - Revised (CYCLE-R) | Baseline and immediately after the intervention (3rd week for the low-intensity arm and 9th week for the high-intensity arm)
  A sentence-to-picture matching tasks that evaluates comprehension of sentences of varying complexity. The scores range from 0 to 100%, with higher scores indicative of better comprehension abilities.
Changes on the Center for Epidemiological Studies Depression Scale (CES-D) | Baseline and immediately after the intervention (3rd week for the low-intensity arm and 9th week for the high-intensity arm)
  The 20-item self-rating questionnaire evaluates perceived mood and level of functioning within the past seven days. The scores range from 0-60. A score equal to or above 16 indicates a person at risk for clinical depression.
Changes on the General Anxiety Disorder scale (GAD-7) | Baseline and immediately after the intervention (3rd week for the low-intensity arm and 9th week for the high-intensity arm)
  The 7-item self-report scale is used to identify anxiety based on problems experienced in the last two weeks. The scores range from 0-21, with higher scores indicative of more pronounced anxiety symptoms.
Changes on the Pittsburgh Sleep Quality Index (PSQI) | Baseline and immediately after the intervention (3rd week for the low-intensity arm and 9th week for the high-intensity arm)
  The self-rating scale used to measure the quality and patterns of sleep. It differentiates "poor" from "good" sleep by measuring seven areas: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction over the last month. The overall score ranges from 0-21, with higher scores indicative of more acute sleep disturbances.
Changes on the Stroke and Aphasia Quality of Life Scale - 39 (SAQOL-39) | Baseline and immediately after the intervention (3rd week for the low-intensity arm and 9th week for the high-intensity arm)
  This questionnaire is specifically designed to assess quality of life in individuals with stroke and aphasia. The overall quality of life score can range from 1 to 5, with higher values indicating better quality of life and overall well-being.
Change on the Modified Rankin Scale (MRS) | Baseline and immediately after the intervention (3rd week for the low-intensity arm and 9th week for the high-intensity arm)
  This is a commonly used 7-point rating scale for measuring the degree of overall disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. MRS is a single item, global outcomes rating scale for patients post-stroke. The measure is scored based on a structured interview. It is used to categorize level of functional independence with reference to pre-stroke activities rather than on observed performance of a specific task. The scale ranges from 0 to 6, with higher scores indicative of more severe disability, with 6 indicating that the patient is dead.
Changes on the National Institute of Health Stroke Scale (NIHSS) | Baseline and immediately after the intervention (3rd week for the low-intensity arm and 9th week for the high-intensity arm)
  This is a widely used clinical scale for measuring impairment in various domains (consciousness, motor, sensory, attention, language) after stroke. It uses a numerical scale to determine stroke severity, health care providers record the person's performance in 11 categories, such as sensory and motor ability. Each domain is rated on a scale from 0 to 2 or 3/4 for certain domains), with 0 indicating no impairment. The total score can range from 0 to 42 points, with higher scores indicating greater severity.
Changes on the Fugl-Meyer Assessment, Upper Extremity portion (FMA-UE) | Baseline and immediately after the intervention (3rd week for the low-intensity arm and 9th week for the high-intensity arm)
  This is a commonly used outcome measure for assessment of sensorimotor recovery after stroke. We will only use the upper extremity portion of the assessment to supplement other study measures focusing on gait and balance. The FMA-UE assesses movement, coordination, and reflexes associated with the shoulder, elbow, forearm, wrist, and hand and is meant to capture stages of motor recovery after stroke. The FMA-UE consists of 33 items with each item scored on a 3-point ordinal scale (0, 1, or 2), with 0 generally corresponding to no function, 1 to partial function, and 2 to perfect function. The items are summed to provide a final score, ranging from 0-66 points, with lower scores indicative of more pronounced motor impairments of the upper extremity.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Ivanova, PhD, Principal Investigator — University of California, Berkeley
Locations (4):
- United States (4):
  - University of California Berkeley, Berkeley, California
  - California State University East Bay, Hayward, California
  - University of San Francisco, San Francisco, California
  - University of California San Francisco, San Francisco, California

IPD SHARING:
Plan to Share IPD: No